CLINICAL TRIAL: NCT05398978
Title: The Effect of e-Registration and mHealth on Institutional Deliveries in the Hazard-prone Areas of Southern Bangladesh: A Protocol for an Open-label Two-arm Non-randomized Controlled Cluster Trial
Brief Title: The Effect of e-Registration and mHealth on Institutional Deliveries in the Hazard-prone Areas
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: North South University (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Ahmed Hossain, Professor, North South University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: NorthSouthU
Record Dates: First submitted 2022-05-23; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Place of Delivery
Keywords: Non-randomized controlled cluster trial; institutional delivery; e-Registration; mHealth
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: The pregnant mothers will be registered in the electronic database, they will be called by the midwives to motivate them for facility delivery and they will receive a text message regarding this.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention arm will be registered in th e-Register database and recieve voice calls and text messages
  Interventions: Other: e-Registration and mHealth
- Control (No Intervention): The control group will be enrolled and followed until their delivery. They will not get the intervention.

INTERVENTIONS:
Other: e-Registration and mHealth — Registration to the electronic database Counseling through voice calls for facility delivery Text messages to promote facility delivery
  Arms: Intervention

SUMMARY:
The study aims to determine the effect of the eRegistration tracking system and mHealth counseling on institutional deliveries to pregnant mothers in the hazard-prone areas of Southern Bangladesh.

DETAILED DESCRIPTION:
The study will be an open-label two-arm non-randomized controlled cluster trial for six months period. Chandpur Sadar, Kachua, and Faridganj sub-districts will be the intervention arm and Bhola Sadar, Charfesson, and Lalmohan sub-districts of the Bhola district will be the control arm. ased system. 28 - 36 weeks of pregnant women will be enrolled, given the intervention, and followed-up until their delivery.

ELIGIBILITY:
Pregnant mothers registered in the FWA register, 19 - 45 years, 28 - 36 weeks pregnant, have access to a mobile phone

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — We will include pregnant mothers for our study. Participant eligibility is based on thier pregnancy status and self-representation of gender identity.
Enrollment: 536 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-11-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of Institutional delivery | 22 weeks
  Normal vaginal deliveries, cesarean sections and assisted vaginal deliveries (forceps and vacuum deliveries) conducted at any healthcare facility by medically trained provider/ skilled birth attendant situated at the study sites will be considered as institutional delivery.
  Numerator: Number of institutional deliveries Denominator: Total deliveries in the study sites (A sum of normal vaginal deliveries, cesarean sections and assisted vaginal deliveries)

SECONDARY OUTCOMES:
Proportion of different mode of deliveries | 22 weeks
  Numerator: Proportion of normal vaginal deliveries, Proportion of cesarean sections, Proportion of forceps and vacuum deliveries Denominator: Total deliveries in the study sites.
Proportion of different birth outcomes | 22 weeks
  Numerator: Proportion of alive babies, Proportion of stillbirths Denominator: Total live births in the study sites.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hossain, Ph.D, MSc, Study Chair — North South University

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data available to other researchers.

REFERENCES:
- [Derived] Chowdhury AT, Jabeen S, Sultana ZZ, Rahman AE, Arifeen SE, Hossain A. Evaluating the impact of e-registration and mHealth on institutional delivery in hazard-prone areas of Bangladesh: A protocol for a non-randomized controlled cluster trial. PLoS One. 2023 Sep 27;18(9):e0271364. doi: 10.1371/journal.pone.0271364. eCollection 2023. PMID 37756321